CLINICAL TRIAL: NCT06006754
Title: Influence of Enteral Microbiome Composition and Microbiome Dependent Metabolites on Mortality of Patients With Cardiogenic Shock
Brief Title: Influence of Enteral Microbiome on Mortality of Patients With Cardiogenic Shock
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Chistos Rammos, Professor Dr. med., University Hospital, Essen
Other Study IDs: Microbiome-Shock-Trial
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock; Microbial Colonization; Out-Of-Hospital Cardiac Arrest; Acute Heart Failure; Acute Myocardial Infarction
MeSH Terms: conditions — Shock, Cardiogenic; Communicable Diseases; Out-of-Hospital Cardiac Arrest | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiogenic shock
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention: observational study

SUMMARY:
Cardiogenic shock is associated with a high mortality. The microbiome is a double-edged sword which can convey protective and detrimental cardiovascular effects. The significance of the enteral micobiome on cardiovascular mortality of patients with cardiogenic shock is still not known.

This study aims to provide a deeper understanding of the role of the enteral microbiome and microbiome dependent metabolites in mortality and disease progression of patients with cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* >18y
* signs of cardiogenic shock regardless of etiology

  * lactate >3mmol/L
  * and signs of organ dysfunction (urine output <30 ml/h, cold extremities, altered mental status)
  * and systolic blood pressure <90 mmHg for >30 minutes or need for vasopressor therapy

Exclusion Criteria:

* pregnancy/lactation period
* antibiotic treatment within >24h
* chronic inflammatory bowel disease
* short bowel syndrome
* artificial bowel outlet
* persistent diarrhea or vomiting in the past 3 months
* simultaneous participation in another interfering nutrition study
* active chemo or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years presenting to the clinic with cardiogenic shock will be included into the study within a 24 hours timeframe after onset
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Correlation between enteral microbiome composition and mortality | Sampling will be performed within 24 hours of onset of cardiogenic shock and clinical evaluation will be performed after 1 month
  Stool samples are collected and clinical evaluation will be performed at below mentioned time points

SECONDARY OUTCOMES:
Correlation between TMAO serum level and mortality | Sampling will be performed within 24 hours of onset of cardiogenic shock and on day 3
  Blood samples are collected at below mentioned time points
Correlation between SCFA serum level and mortality | Sampling will be performed within 24 hours of onset of cardiogenic shock and on day 3
  Blood samples are collected at below mentioned time points
Correlation between inflammatory profile (CRP, PCT, Interleukin panel) and mortality | Sampling will be performed within 24 hours of onset of cardiogenic shock and on day 3
  Blood samples are collected at below mentioned time points

CONTACTS AND LOCATIONS:
Overall Officials: Christos Rammos, Prof. Dr., Study Chair — University Clinic Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No